CLINICAL TRIAL: NCT01208428
Title: Cognitive Behavioral Treatments for Depression in Patients With Chronic Illness
Brief Title: Cognitive Behavioral Treatments for Depression in Chronic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00026533
Record Dates: First submitted 2010-09-22; First posted 2010-09-24 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Major Depression
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional cognitive behavioral therapy (Active Comparator): Subjects randomized to this arm will receive conventional cognitive behavioral therapy for the treatment of major depression
  Interventions: Behavioral: Conventional cognitive behavioral therapy
- Religious cognitive behavioral therapy (Experimental): Subjects randomized to this arm will receive conventional cognitive behavioral therapy, but their religious beliefs will be utilized as a resource in the therapy
  Interventions: Behavioral: Religious cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Conventional cognitive behavioral therapy — Conventional cognitive behavioral therapy is a standard treatment for depression. There will be ten 50-minute sessions delivered.
  Arms: Conventional cognitive behavioral therapy
Behavioral: Religious cognitive behavioral therapy — Religious cognitive behavioral therapy is conventional cognitive behavioral therapy that includes consideration of the patient's religious beliefs in therapy. Subjects will receive ten 50-min sessions of therapy
  Arms: Religious cognitive behavioral therapy

SUMMARY:
Duke University Medical Center in collaboration with Glendale Adventist Medical Center propose a randomized clinical trial of conventional cognitive behavior therapy (CCBT) vs. religious cognitive behavior therapy (RCBT) for major depression in medical patients with chronic disabling illness. Therapists will deliver the treatment in real time over the Internet and/or by telephone to increase treatment access. This planning grant seeks support for a two-site study (North Carolina and California) that consists of two phases. In Phase I (Rounsaville 1a) the investigators will conduct an open trial of 30 patients to assess subject recruitment, refine RCBT and CCBT manuals and protocol, assess compliance with treatment, acceptability of treatment and delivery system (online vs. telephone), and allow therapists gain experience with delivery system and RCBT.

In Phase II (Rounsaville 1b) the investigators will conduct a randomized proof of concept comparison of CCBT vs. RCBT that will demonstrate feasibility and confirm the expected clinically meaningful difference for a definitive R01 application. In Phase II, 70 religious patients ages 18-85 with a new episode of major depression (MINI), scores of 16-35 on the Beck Depression Inventory (BDI), and at least one chronic disabling medical illness will be randomized to either CCBT or RCBT. The trial will consist of ten 50 min sessions administered by master's level therapists and delivered over 12 weeks. The primary endpoint will be BDI score at baseline, 4, 8, 12, and 24-week follow-up. Christian, Jewish, Hindu, Buddhist, and Muslim versions of the RCBT manual will be developed, and CBT experts in each of these traditions will supervise therapists delivering the intervention to patients from these faith traditions.

The purpose of this study is to determine feasibility and effect sizes for a future, fully powered treatment study. The importance is that results will be relevant to therapists well beyond those who explicitly practice pastoral counseling, extending to many secular therapists as well. If 65% of Americans indicate that religion is an important part of daily life and the vast majority of chronically ill medical patients wish to include it in their therapy, then all therapists (whether they have explicit training in pastoral counseling or not) are likely to encounter patients in which this approach would be applicable.

ELIGIBILITY:
Inclusion Criteria:

* chronic disabling medical illness
* religion at least somewhat important to patient
* major depressive disorder by MINI neuropsychiatric interview
* Beck Depression Inventory scores of 16-28 (moderately severe depression)
* live near Durham, North Carolina, or near Glendale, in Southern California

Exclusion Criteria:

* significant cognitive impairment
* significant suicidal thoughts or risk
* no access to telephone

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | Baseline
  Quantitative assessment of depressive symptoms
Beck Depression Inventory | 4 weeks
  Quantitative assessment of depressive symptoms
Beck Depression Inventory | 8 weeks
  Quantitative assessment of depressive symptoms
Beck Depression Inventory | 12 weeks
  Quantitative assessment of depressive symptoms
Beck Depression Inventory | 24 weeks
  Quantitative assessment of depressive symptoms

SECONDARY OUTCOMES:
Duke Social Support Index (abbreviated) | Baseline
  Measures amount of social support and satisfaction with it.
Duke Social Support Index (abbreviated) | 12 weeks
  Measures amount of social support and satisfaction with it
Duke Social Support Index | 24 weeks
  Measures amount of social support and satisfaction with it.

CONTACTS AND LOCATIONS:
Overall Officials: Harold G Koenig, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Glendale Adventist Medical Center, Glendale, California
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Propst LR, Ostrom R, Watkins P, Dean T, Mashburn D. Comparative efficacy of religious and nonreligious cognitive-behavioral therapy for the treatment of clinical depression in religious individuals. J Consult Clin Psychol. 1992 Feb;60(1):94-103. doi: 10.1037//0022-006x.60.1.94. PMID 1556292
- [Background] Koenig HG. Religion and remission of depression in medical inpatients with heart failure/pulmonary disease. J Nerv Ment Dis. 2007 May;195(5):389-95. doi: 10.1097/NMD.0b013e31802f58e3. PMID 17502804
- [Background] Koenig HG, George LK, Peterson BL. Religiosity and remission of depression in medically ill older patients. Am J Psychiatry. 1998 Apr;155(4):536-42. doi: 10.1176/ajp.155.4.536. PMID 9546001